CLINICAL TRIAL: NCT01524237
Title: Biomarker Study: Impact of Single Doses of LY2979165 and LY2140023 on the Ketamine-Challenge Pharmacological MRI Assay in Healthy Male Subjects
Brief Title: A Study of LY2979165 and LY2140023 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 13882; I4S-EW-HHCC (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — LY 2140023; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 10 mg LY2140023 + ketamine (Experimental): Single oral dose of 10 mg LY2140023 followed by intravenous (IV) ketamine during one of the crossover periods
  Interventions: Drug: LY2140023; Other: Ketamine
- 20 mg LY2979165 + ketamine (Experimental): Single oral dose of 20 mg LY2979165 followed by IV ketamine during one of the crossover periods
  Interventions: Drug: LY2979165; Other: Ketamine
- 40 mg LY2140023 + ketamine (Experimental): Single oral dose of 40 mg LY2140023 followed by IV ketamine during one of the crossover periods
  Interventions: Drug: LY2140023; Other: Ketamine
- 60 mg LY2979165 + ketamine (Experimental): Single oral dose of 60 mg LY2979165 followed by IV ketamine during one of the crossover periods
  Interventions: Drug: LY2979165; Other: Ketamine
- 160 mg LY2140023 + ketamine (Experimental): Single oral dose of 160 mg of LY2140023 followed by IV ketamine during one of the crossover periods
  Interventions: Drug: LY2140023; Other: Ketamine
- Placebo capsules + ketamine (Placebo Comparator): Single oral dose of placebo capsules followed by IV ketamine during one of the crossover periods
  Interventions: Other: Placebo; Other: Ketamine
- Placebo tablets + ketamine (Placebo Comparator): Single oral dose of placebo tablets followed by IV ketamine during one of the crossover periods
  Interventions: Other: Placebo; Other: Ketamine

INTERVENTIONS:
Drug: LY2979165 — Capsules administered orally
  Arms: 20 mg LY2979165 + ketamine; 60 mg LY2979165 + ketamine
Drug: LY2140023 — Tablets administered orally
  Arms: 10 mg LY2140023 + ketamine; 160 mg LY2140023 + ketamine; 40 mg LY2140023 + ketamine
Other: Placebo — Administered orally
  Arms: Placebo capsules + ketamine; Placebo tablets + ketamine
Other: Ketamine — Administered intravenously (IV)

SUMMARY:
This study will be comprised of 2 parts, Part A and Part B, both in healthy male participants.

Part A of the study will investigate the safety of intravenous (IV) ketamine administration after single oral doses of LY2979165 (capsules) or LY2140023 (tablets). Part A will be completed before starting Part B.

Part B of this study will investigate whether different dose levels of LY2979165 or LY2140023, when administered before ketamine, result in changes to the images on a brain scan seen with ketamine alone. Brain imaging is currently used for a number of reasons including understanding where in the brain medicines have their effects. Ketamine is an anesthetic used in this study to activate particular regions of the brain.

The single oral doses of LY2979165 to be used in both parts of the study are 20 and 60 mg with matching dummy drug (placebo) for each dose.

The doses for LY2140023 are 10, 40, and 160 mg with matching placebo for each dose.

Screening is required within 28 days prior to the start of the study and follow up 7-14 days after the last dose of study drug. The study will last up to 8-weeks for an individual participant.

ELIGIBILITY:
Inclusion Criteria:

* are overtly healthy, right-handed, Caucasian (non-Hispanic White by self report) males, as determined by medical history and physical examination
* agree to use an effective method of birth control during the study and for a period of 3 months after the final dose of study drug
* if female partners are of child-bearing potential, agree to use 2 effective methods of birth control during the study and for a period of 3 months after the final dose of study drug

  * one (1) of these methods must be a male or female condom used in conjunction with spermicidal gel, foam, cream, film or suppository
  * the other method can be any of the following:

    * diaphragm or cervical vault cap used in conjunction with spermicidal gel, foam, cream, film, or suppository
    * male partner sterilization
    * true abstinence (which is in line with the participant's usual lifestyle choice; withdrawal or calendar methods are not considered acceptable)
    * placement of an effective intrauterine device (IUD) (Consideration should be given to the type of device or system being used, as there are higher failure rates quoted for certain types)
    * established use of oral, injected, or implanted hormonal methods of contraception
* have a body mass index (BMI) of 18.0 to 30.0 kg/m^2, inclusive, and weigh 50.0 to 100.0 kg, at the time of screening
* have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* have venous access sufficient to allow for blood sampling and administration of intravenous (IV) ketamine as per the protocol
* are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site

Exclusion Criteria:

* are currently enrolled in, have completed or discontinued within the last 90 days from, a clinical trial involving an investigational product; or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* have known allergies to LY2979165, LY2140023, ketamine, related compounds or any components of the formulations
* are persons who have previously completed or withdrawn from this study or any other study investigating LY2979165 or LY2140023
* have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study or have a PR interval greater than 200 msec, or QTc interval greater than 450 msec
* have an abnormal resting, supine blood pressure (BP), defined as systolic blood pressure (BP) greater than 150 mm Hg or diastolic BP greater than 85 mm Hg, or a heart rate (HR) outside the range of 40 to 85 beats per minute (bpm), inclusive
* have a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data
* have a history of or regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* show evidence of significant active neuropsychiatric disease, suicidal risk (including suicidal ideation as assessed by the Columbia Suicide Severity Rating Scale [C-SSRS]) or have a first degree relative with a history of psychosis
* show evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies
* show evidence of hepatitis C and/or positive hepatitis C antibody
* show evidence of hepatitis B and/or positive hepatitis B surface antigen
* have used or intend to use over-the-counter or prescription medication within 7 days prior to dosing. Herbal supplements must be discontinued 28 days prior to the first dose of trial medication. At the discretion of the investigator a shorter drug free or discontinuation period may be acceptable depending on the precise drugs/supplements taken. As an exception, paracetamol or acetaminophen may be used at doses of up to 1 g/day
* have donated blood of more than 500 mL within the last month
* have an average weekly alcohol intake that exceeds 28 units per week, or are unwilling to stop alcohol consumption for 48 hours prior to dosing until the completion of each study period and restrict consumption to no more than 3 units per day for the duration of the study (1 unit = 190 mL of beer; 87.5 mL of wine; 25 mL of distilled spirits)
* use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day or unable/unwilling to abide by the clinical research unit (CRU) smoking restrictions from admission to the CRU until discharge for each study period
* consume caffeine equivalent to more than 6 cups of coffee per day, on a habitual basis, or are unable to abide by the study restrictions for caffeine/xanthine use (that is, refrain from consuming caffeine/xanthine-containing drinks and foods (such as coffee, tea, cola, and chocolate) from admission to the CRU until discharge for each study period
* in the opinion of the investigator or sponsor, are unsuitable for inclusion in the study
* Have increased risk of seizures as evidenced by a history of more than 1 seizure (except childhood febrile seizure), history of electroencephalogram (EEG) with epileptiform activity, history of stroke; surgery to the cerebral cortex; or head trauma with loss of consciousness

Additional criteria for Part B only:

* History of claustrophobia or inability to tolerate mock scanner environment during habituation/screening session
* Fulfillment of any of the magnetic resonance imaging (MRI) contraindications on the standard radiography screening questionnaire (for example, history of surgery involving metal implants)

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Part A: Number of participants with one or more drug related adverse events (AEs) or any serious AEs | Part A: Day 1 through 3
Part B: Changes in hemoglobin oxygenation in the brain during ketamine infusion | Part B: Day 1

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration curve (AUC) of LY2979165, LY2140023, and active metabolites | Up to Day 3
Pharmacokinetics: Maximum concentration (Cmax) of LY2979165, LY2140023, and active metabolites | Up to Day 3
Pharmacokinetics: Area under the concentration curve (AUC) of ketamine and nor-ketamine | Up to Day 3
Relationship between active compounds' exposure (e.g. AUC) and hemoglobin oxygenation in the brain | Part B: Up to 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Greater London
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, UK